CLINICAL TRIAL: NCT04244565
Title: Effect of Self-Directed Versus Traditional Clinical Learning Model on Nurses' Airway Management Competencies and Patients' Airway Related Incidents
Brief Title: Self-Directed Versus Traditional Clinical Learning Model on Nurses' Airway Management Competencies
Acronym: SDLMvsTCLM
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Elhabashy, Lecturer, Cairo University
Other Study IDs: FWA00019803
Record Dates: First submitted 2020-01-07; First posted 2020-01-28 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Airway Morbidity; Nurse's Role; Airway Obstruction; Nurse's Scope of Practice
Keywords: Self-directed, Traditional Clinical Learning
MeSH Terms: conditions — Airway Obstruction | interventions — Nurses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Self-directed clinical learning: examining the effect of Self-directed clinical learning model as compared to the traditional models to improve nurses' Airway management competencies and minimize airway related incidents.
  Interventions: Behavioral: Self-directed model of clinical learning for nurses

INTERVENTIONS:
Behavioral: Self-directed model of clinical learning for nurses — the instructors play a facilitating role while, learners actively participate in identifying their own learning needs, learning goals, allocating resources & decide whether learning method can be used, and engaging in self-reflection & evaluation.
  Other Names: compared to the traditional models

SUMMARY:
Effect of Self-Directed Versus Traditional Clinical Learning Model on Nurses' Airway Management Competencies and Patients' Airway Related Incidents

Introduction Airway crisis situations in ICUs (Intensive Care Units) are common, complex, dynamic and time-sensitive contexts, that pose a significant threat to patient safety, and are a major source of preventable errors. Airway management has the highest priority in patient care, it is the first step in the (ABCDE) approach. The concept of Airway management in nursing perspective includes any nursing procedures and techniques required to keep the airway open and prevent aspiration. Adult learning is a practice in which adults engage in systematic and sustained learning activities in order to gain new forms of knowledge, skills or values. Most adult education is voluntary; therefore, the participants are generally self-motivated. Continuing education (CE) of nurses is increasingly necessary to keep abreast of rapid changes in patient care due to advancements in knowledge and technology and improve their ability to serve the patients safely. Although nursing care has been changed significantly over the past 30 years, methods for clinical training nurses have not. A popular or traditional model for clinical teaching of nurses, including but not limited to; integrating lectures, skills laboratory training and supervised clinical experience. A benefit of this model is the opportunity to assist nurses to integrate the concept learned in class or skill lab in patient care. Also, the instructor can select clinical activities that best meet nurses' needs and are consistent with hospital goals. While, Self-directed learning (SDL) is one of modern approaches of clinical learning, the concept of SDL originates from the Adult Learning Theory, it is a process in which the instructors play a facilitating role while, learners actively participate in identifying their own learning needs, learning goals, allocating resources & decide whether learning method can be used, and engaging in self-reflection & evaluation. The positive outcomes of SDL including but not limited to, greater self-control, self-confidence, autonomy, and lifelong learning skills. In essence the aim of this study will be examining the effect of Self-directed clinical learning model as compared to the traditional models to improve nurses' Airway management competencies and minimize airway related incidents.

Research Hypothesis H1: Critically care nurses who will approach self-directed clinical learning model (μ1) will have a higher level of Airway management skills (μ2), (H1: μ1 > μ2).

H1: Intensive care units who will approach self-directed clinical learning model to learn their working nurses (μ1) will have a lower frequency of patients' airway-related incidents (μ2), (H1: μ1 < μ2).

Subjects and Methods True experimental, prospective, and comparative research design will be utilized in the current study. This study will be conducted at selected two Adult Intensive Care Units, A convenience sample of 60 male and female Critically Care Nurses who are working in the selected Intensive Care Unit, will be recruited to the study. The sample size estimated by (G Power analysis) (independent t tests - One tail, Effect size = 0.65, α = 0.05, Power (1-β) = 0.80, balanced allocation ratio 1:1). The total sample size will be divided into two groups (study and control). All nurses should be corresponded to specific inclusion criteria.

Five tools will be formulated to collect data pertinent to the study.

Procedure The study will be conducted through three phases; preparation & designation, implementation, and follow up & evaluation phase. The 1st Part will be initiated by allocating the selected ICUs randomly into two paired settings, one for applying traditional learning (control ICU) and the other for self-directed learning experimentation (study ICU). the nurses who are working in selected ICUs and correspond to the inclusion criteria, will be randomly distributed into two equal groups (30 nurses in each group). The nurses who are working in study ICU will be asked to fill out the nurses' readiness assessment sheet to learn independently. The nurses who will demonstrate a high readiness score (>80%) for independent learning will be included. Once implantation is complete, the follow-up and evaluation phase will be initiated by daily monitoring of the occurrence of patients' airway related incidents in both control and study ICUs for a continuous three months. Then, the nurses' knowledge and practices (in the control group) will be evaluated two times, 1st time will be 1 month after the implementation phase, and the second time will be after 3 months from the 1st evaluation (to measure the retention of given education and training). Upon completion of data collection, descriptive and inferential statistics will be utilized to test for differences among the study and control group subjects.

DETAILED DESCRIPTION:
Effect of Self-Directed Versus Traditional Clinical Learning Model on Nurses' Airway Management Competencies and Patients' Airway Related Incidents

Introduction

Airway crisis situations in ICUs (Intensive Care Units) are common, complex, dynamic and time-sensitive contexts, that pose a significant threat to patient safety, and are a major source of preventable errors [1]. Although, only a few studies have demonstrated the airway incidents in ICUs, 7.04% of ICU patients developed airway incidents [2]. The UK National Reporting and Learning Centre identified that 82% of ICU airway incidents occurred in patient with ETT, with 25% contributing to the patient's death [3]. The concept of Airway management in nursing perspective includes any nursing procedures and techniques required to keep the airway open and prevent aspiration [4]. In fact, Airway management has the highest priority in patient care, it is the first step in the (ABCDE) approach. Several nursing related factors that can directly or indirectly cause a patient to have airway crises either patient intubated or even non-intubated, such factors include a partial or complete airway obstruction, injury or infection [5,6]. However, Airway management procedures and techniques (Table 1) are rapidly changing, there is a need for structured innovative training models related to Airway management education for critical care nurses to develop nurses' competences and subsequently will enhance patients' outcomes [7,8,9].

Adult learning has speciﬁc characteristics, adult education is a practice in which adults engage in systematic and sustained learning activities in order to gain new forms of knowledge, skills or values. Adults have already accumulated knowledge and work experience which can add to their learning experience. Most adult education is voluntary; therefore, the participants are generally self-motivated. Furthermore, adults apply their knowledge in a practical fashion to learn effectively. They must have a reasonable expectation that the knowledge they gain will indeed help them further their goals [10].

Continuing education (CE) of nurses is increasingly necessary to keep abreast of rapid changes in patient care due to advancements in knowledge and technology, nurses also should be well motivated to enroll in CE hospital activity to upgrade their professional skills and knowledge to remain current in their professional practices and improve their ability to serve the patients safely [11]. Clinical placements provide opportunities for nurses to learn experientially. To create a constructive learning environment nursing staff, need to be friendly, approachable, available and willing to learn. Also, CE should be providing adequate opportunities for nurses to develop conﬁdence and competence in clinical skill with a focus on nurses' learning needs rather than service needs of the facilities [12].

Although nursing care has been changed significantly over the past 30 years, methods for clinical training nurses have not [13]. A popular or traditional model for clinical teaching of nurses, including but not limited to; integrating lectures, skills laboratory training and supervised clinical experience. A benefit of this model is the opportunity to assist nurses to integrate the concept learned in class or skill lab in patient care. Also, the instructor can select clinical activities that best meet nurses' needs and are consistent with hospital goals [14]. In addition, the low confidant nurses prefer this type of clinical teaching because they feel more secure [15]. On the other side, the traditional model for clinical teaching contributes to poor critical thinking and reasoning development among nurses and results in task-oriented approaches to teaching and learning. Consequently, nurses may lack the capacity to think through interventions that lead to positive patient outcomes [16]. Therefore, there is a need to find innovative approaches to effectively train nurses to better prepare them for today's health care environment. These innovative approaches may increase the effectiveness and efficiency of the clinical nursing education system [13].

Self-directed learning (SDL) is one of these modern approaches of clinical learning, the concept of SDL originates from the Adult Learning Theory. This theory suggests that adults are pragmatic and problem-focused individuals whose learning are mainly affected by experiential rather than passive approaches [17]. Self-directed learning was applied and examined on nursing students as well as working nurses who are engaged in an on-going continuing training [18]. Self-directed learning is a process in which the instructors play a facilitating role while, learners actively participate in identifying their own learning needs, learning goals, allocating resources & decide whether learning method can be used, and engaging in self-reflection & evaluation. The positive outcomes of SDL including but not limited to, greater self-control, self-confidence, autonomy, and lifelong learning skills [17]. While, SDL may helpful, there is an increasing awareness that SDL is not universally applicable to all learners and all situations. Also, the majority of nurses not familiar with SDL approach of learning they preferred and felt more secure with traditional teacher-centered approach as they usually learned in schools [19]. Self-directed learning can be challenging, even for the brightest and most motivated nurses. Therefore, it should apply in a systematic way to maximize the benefits. four key stages to apply SDL; being ready to learn independently, setting learning goals, engaging in the learning process by understanding themselves and their needs (the discrepancy between the present level of competence and the required level of competency), and evaluating learning [20, 21].

Successful independent study requires certain responsibilities or roles of both nurses and instructor. It is useful for both to communicate as to whether each feels the other is fulfilling their share of the responsibility. nurses' roles include; self-assess readiness to learn, define your learning goals, monitor learning process, be self-motivated, re-evaluate and alter goals as required, consult with instructor as required. While, instructors' roles; Build a co-operative learning environment, help to motivate and direct the nurses' learning experience, facilitate learning, be available for consultations as appropriate during the learning process, serve as an advisor rather than a formal instructor [22]. In essence the aim of this study will be examining the effect of Self-directed clinical learning model as compared to the traditional models to improve nurses' Airway management competencies and minimize airway related incidents.

Research Hypothesis H1: Critically care nurses who will approach self-directed clinical learning model (μ1) will have a higher level of Airway management skills (μ2), (H1: μ1 > μ2).

H1: Intensive care units who will approach self-directed clinical learning model to learn their working nurses (μ1) will have a lower frequency of patients' airway-related incidents (μ2), (H1: μ1 < μ2).

Subjects and Methods

Research Design:

True experimental, prospective, and comparative research design will be utilized in the current study. The study will be conducting a nursing self-directed clinical learning model as compared to the traditional models to improve nurses' Airway management competencies and minimize patients' airway related incidents.

Ethical Consideration:

An official permission to conduct the proposed study will be obtained from the ethical committee. Also. Participation in the study is voluntary; each subject has the right to withdraw from the study when he or she wants. Informed consent will be obtained from the subjects. Confidentiality and anonymity of the subjects are assured through coding of all data; subjects will be assured that these data will not be reused in another research without their permission, collected data will be used for the purpose of the research only and The entire needed sample in the study will be followed until been analyzed. All information taken will be protected and will not affect their annual appraisal by any mean. The formulated database and the result of the current study will be raising the awareness of all health professionals and incorporating in the future plan of care.

Procedure:

The study will be conducted through three phases; preparation & designation, implementation, and follow up & evaluation phase. The preparation & designation phase will be concerned with taken the official permission and ethical approval. Also, it includes a recent review of related literatures, and preparation of the different (constructed and adapted) study tools and formulate the latest evidenced educational content and materials related to airway nursing management. These tools and educational content will be revised by medical and nursing expert to ensure its content validity.

Once the official permission and ethical approval are granted to proceed the proposed study, the implementation phase will be applied in two parts:

The 1st Part will be initiated by allocating the selected ICUs randomly into two paired settings, one for applying traditional learning (control ICU) and the other for self-directed learning experimentation (study ICU). the nurses who are working in selected ICUs and correspond to the inclusion criteria, will be randomly distributed into two equal groups (30 nurses in each group). The nurses who are working in study ICU will be asked to fill out the nurses' readiness assessment sheet to learn independently (tool 4). The nurses who will demonstrate a high readiness score (>80%) for independent learning will be included. if the nurses number exceeding the intended number (30 nurses), the highest scores will be selected.

Self-directed clinical learning model:

The concept of Airway management will be nominated for participant nurses to be an area of investigation. each nurse will be asked to fulfill the pre-structured Learning contract between nurses and instructors within one week, the contract will include the following items.

* Goals for the area of learning (the researcher will confirm the congruence with the expected goals).
* Structure and sequence of activities.
* Timeline for completion of activities (maximum one month).
* Details about resource materials for each goal.
* Feedback and evaluation as each goal is completed.
* Meeting plan with the instructors.
* Self-reflection and self-evaluation methods. the researchers will facilitate all nurses' stated resources incorporation with hospital manager such as (Sill lab., computer lab., internet, hard books, digital books, clinical instructions, or Egyptian Knowledge Bank).

Traditional clinical learning model It will concern the Airway management competencies; it will be given within one month and it will take place during working hours.

1. the researcher will divide the participant (30 nurses) into two main groups (15 nurses in each), each group will be given pre-scheduled integrated lectures related to theoretical background of Airway management. Four lectures will be given once per-week, 2 hours long, written handouts will be given.
2. After each driven lecture, the researcher will give a supportive four hours skill laboratory training by traditional 2 stages, methods ("see one, do one"). This traditional "2-stage approach" was standard for improving clinical practices.
3. Then, the researchers will provide a clinical supervision and guidance for the participant nurses to ensure that they will able to apply what they learned in real settings.

Once implantation is complete, the follow-up and evaluation phase will be initiated by daily monitoring of the occurrence of patients' airway related incidents in both control and study ICUs for a continuous three months (tool 3). Then, the nurses' knowledge and practices (in the control group) will be evaluated two times, 1st time will be 1 month after the implementation phase, and the second time will be after 3 months from the 1st evaluation (to measure the retention of given education and training), tools (1, 2) will be utilized, and it will be completed by blinded assessors (who were not part of the research team). On the other side, the study group of self-directed learning will be self-evaluated by using tools (1, 2) and also will be evaluated two times like control group. Finally, the researcher will compare the results (outcome given by self-directed learning) to the collected baseline data (control group) which will be given as usual ongoing traditional learning.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in this study.
* Working for at least one month in the current position.
* Maximum two years of experience in critical care.

Exclusion Criteria:

* Nurses who attended any educational courses in Airway management in last 6 months, will be excluded.
* Nurses planning to leave work 6 months later, will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A convenience sample of 60 male and female Critically Care Nurses who are working in the selected Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Structured questionnaire schedule to assess nurses' knowledge (Level) regarding Airway management related issues. | 5 months
  Nurses' Airway management competencies need a wide theoretical background aimed to practice based on rational and evidence. Airway management has the highest priority in patient care. Nurses' knowledge regarding Airway management consists of different issues such as; (1) Causes of Airway obstructions (2) Ways to maintain Airway clear (3) Management of ETT cuff pressure. (4) Airway assessment items. This questionnaire will be self-administrated for the group who will be applied self-directed clinical learning model. While, it will be conducted by the clinical instructor by interview for the group who will be applying the traditional clinical learning model. The tool consists of 20 MCQ questions, each right answer will be given one score, total scores will be 20 grades. Those who obtained > 80% will be considered as having a satisfactory knowledge level.
Structured observational checklist to monitor the nurses' practices (Level) regarding Airway management skills | 3 months
  Nurses' Airway management skills include different nursing procedures or maneuvers aimed to maintain airway clear. Airway management has the highest priority in patient care. Nurses' airway management skills such as; (1) Suction to remove secretion (2) Airway maneuvers e.g. head-tilt and chin-lift (3) Proper fixation and care of ETT (4) Management of ETT cuff pressure (5) Oral care (6) Airway assessment skills. This tool will be self-administrated for the group who will be applied self-directed clinical learning model. While, it will be conducted by the clinical instructor by direct observation for the group who will be applying the traditional clinical learning model. The tool consists of 50 items, each item checked as; done complete and correct was given two scores, done incomplete was given one score, and not done or done incorrect was given zero, eventually, those who obtained > 80% will be considered as having a satisfactory practical level.
Patients' Airway Related Incidents (Rate) | 3 months
  Patients' airway related Incidents defined as any airway safety problems or events for either intubated or non-intubated patients, which led to partial or complete airway obstruction, injury or infection. Such as; accumulation of secretion, aspiration or edema. the researcher will be assessed the incidents by pre-structured Patients' airway related Incidents assessment checklist which collect and categorize the incidents (events) within the planned time frame.

OTHER OUTCOMES:
Nurses' Readiness to Learn Independently (Rate) | 1 month
  Evaluation of participant nurses' readiness to learn independently is very important before assign the participant nurses to the study or control group of the current study. This tool will be completed by the nurse herself in addition to receive peer feedback. Nurses' readiness to learn independently assessment questionnaire will be the utilized tool. According to this tool's score the participant nurses will be recruited in either the group who will apply the traditional clinical learning model (control group) or the group of nurses who demonstrate the highest score will apply self-directed clinical learning model (study group).

CONTACTS AND LOCATIONS:
Overall Officials: Gaber, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nguyen LHP, Bank I, Fisher R, Mascarella M, Young M. Managing the airway catastrophe: longitudinal simulation-based curriculum to teach airway management. J Otolaryngol Head Neck Surg. 2019 Feb 19;48(1):10. doi: 10.1186/s40463-019-0332-0. PMID 30782200
- [Background] Chatterjee, A., Islam, S., & Divatia, J. V. (2004). Airway accidents in an intensive care unit.
- [Background] Higgs A, Cook TM, McGrath BA. Airway management in the critically ill: the same, but different. Br J Anaesth. 2016 Sep;117 Suppl 1:i5-i9. doi: 10.1093/bja/aew055. Epub 2016 May 4. No abstract available. PMID 27147544
- [Background] da Silva LFM, Pascoal LM, Nunes SFL, de Sousa Freire VEC, de Araujo Almeida AG, Gontijo PVC, Neto MS. Ineffective Airway Clearance in Surgical Patients: Evaluation of Nursing Interventions and Outcomes. Int J Nurs Knowl. 2019 Oct;30(4):251-256. doi: 10.1111/2047-3095.12242. Epub 2019 Mar 27. PMID 30916452
- [Background] Divatia, J. V., & Bhowmick, K. (2005). Complications of endotracheal intubation and other airway management procedures. Indian J Anaesth, 49(4), 308-18
- [Background] Holbery, N., & Newcombe, P. (2016). Emergency nursing at a glance. John Wiley & Sons.
- [Background] Huitink, J. M., & Bretschneider, J. H. (2015). Airway Management Academy: A global initiative to increase patient safety during airway management by medical education. Trends in Anaesthesia and Critical Care, 5(1), 42-47
- [Background] Spaliaras, J., Streiff, A., Mann, G., & Straker, T. (2019). Teaching and training in airway management: Time to evaluate the current model?. Airway, 2(1), 28
- [Background] Lindkaer Jensen NH, Cook TM, Kelly FE. A national survey of practical airway training in UK anaesthetic departments. Time for a national policy? Anaesthesia. 2016 Nov;71(11):1273-1279. doi: 10.1111/anae.13567. Epub 2016 Sep 28. PMID 27679501
- [Background] Ni C, Hua Y, Shao P, Wallen GR, Xu S, Li L. Continuing education among Chinese nurses: a general hospital-based study. Nurse Educ Today. 2014 Apr;34(4):592-7. doi: 10.1016/j.nedt.2013.07.013. Epub 2013 Aug 7. PMID 23931929
- [Background] Croxon L, Maginnis C. Evaluation of clinical teaching models for nursing practice. Nurse Educ Pract. 2009 Jul;9(4):236-43. doi: 10.1016/j.nepr.2008.06.004. Epub 2008 Aug 21. PMID 18722161
- [Background] Niederhauser V, Schoessler M, Gubrud-Howe PM, Magnussen L, Codier E. Creating innovative models of clinical nursing education. J Nurs Educ. 2012 Nov;51(11):603-8. doi: 10.3928/01484834-20121011-02. Epub 2012 Oct 11. PMID 23061436
- [Background] Shellenbarger, T., Gaberson, K., & Oermann, M. (2018). Clinical teaching strategies in nursing. Springer publishing company.5th ed
- [Background] Luhanga, F. L. (2018). Learning in the traditional-faculty supervised teaching model: part 1-the nursing students' perspective. J Nurs Educ Pract, 8, 89-102
- [Background] Hill, L., & Williams, E. P. (2017). Contemporary Models for Clinical Nursing Education
- [Background] Ghiyasvandian S, Malekian M, Cheraghi MA. Iranian Clinical Nurses' Activities for Self-Directed Learning: A Qualitative Study. Glob J Health Sci. 2015 Sep 1;8(5):48-58. doi: 10.5539/gjhs.v8n5p48. PMID 26652072
- [Background] Montin, L., & Koivisto, J. M. (2014). Effectiveness of self-directed learning methods compared with other learning methods in nursing education related to nursing students' or registered nurses' learning outcomes: a systematic review protocol. JBI Database of Systematic Reviews and Implementation Reports, 12(2), 1-8
- [Background] Levett-Jones TL. Self-directed learning: implications and limitations for undergraduate nursing education. Nurse Educ Today. 2005 Jul;25(5):363-8. doi: 10.1016/j.nedt.2005.03.003. PMID 15894411
- [Background] Kim, R., Olfman, L., Ryan, T., & Eryilmaz, E. (2014). Leveraging a personalized system to improve self-directed learning in online educational environments. Computers & Education, 70, 150-160
- [Background] Murad MH, Varkey P. Self-directed learning in health professions education. Ann Acad Med Singap. 2008 Jul;37(7):580-90. PMID 18695772
- [Background] Self-Directed Learning: A Four-Step Process. University of Waterloo. (2019, March 4). Retrieved April 12, 2019, from https://uwaterloo.ca/centre-for-teaching-excellence/teaching-resources/teaching-tips/tips-students/self-directed-learning/self-directed-learning-four-step-process
- [Background] Manning, G. (2007). Self-directed learning: A key component of adult learning theory. Business and Public Administration Studies, 2(2), 104
- [Background] Terry, A. (2017). Clinical research for the doctor of nursing practice. (3rd ed). Jones & Bartlett Publishers
- [Derived] Elhabashy S, Moawad A. Effect of self-directed versus traditional learning model on nurses' airway management competencies and patients' airway-related incidents. BMC Nurs. 2024 Aug 27;23(1):599. doi: 10.1186/s12912-024-02232-0. PMID 39192309